CLINICAL TRIAL: NCT05228912
Title: Analysis of Immunization Time, Amplitude and Adverse Events of 7 Different Vaccines Against SARS-COV-2 Across 4 Countries
Brief Title: Immunization of 7 Different Vaccines Against SARS-COV-2 Across 4 Countries.
Status: Completed | Type: Observational
Sponsor: Hospital Clinica Nova (Other)
Collaborators: Universidad de Monterrey (Other); Politecnico di Milano (Other); Hospital de San Jose (Other); Hospital Interzonal de Agudos San Juan Bautista (Other); Federal University of Minas Gerais (Other); Fundación San Francisco Javier (Unknown); Humanitas Research Hospital IRCCS, Rozzano-Milan (Other)
Responsible Party: Principal Investigator, Maria Elena Romero Ibarguengoitia, MD, MS, PHD, Hospital Clinica Nova
Other Study IDs: 7 vaccines against COVID-19
Record Dates: First submitted 2022-02-04; First posted 2022-02-08 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Vaccine Adverse Reaction; COVID-19; Vaccine Reaction
Keywords: COVID-19; immune response; Adverse reaction
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — plasma samples to determine the amount of specific anti-S1 and anti-S2 IgG antibodies against SARS-CoV-2 in
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- BNT162b2 mRNA: Group of patients of any age, any sex, that will receive a complete scheme of approved BNT162b2 mRNA vaccination , assigned by a local government vaccination campaign. It can also include patients that receive a third or fourth boost.
  Interventions: Drug: COVID-19 Vaccines
- mRNA-1273: Group of patients of any age, any sex, that will receive a complete scheme of approved mRNA-1273 vaccination, assigned by a local government vaccination campaign. It can also include patients that receive a third or fourth boost.
  Interventions: Drug: COVID-19 Vaccines
- ChAdOx1-S: Group of patients of any age, any sex, that will receive a complete scheme of approved ChAdOx1-S vaccination, assigned by a local government vaccination campaign. It can also include patients that receive a third or fourth boost.
  Interventions: Drug: COVID-19 Vaccines
- Ad26.COV2: Group of patients of any age, any sex, that will receive a complete scheme of approved Ad26.COV2 vaccination, assigned by a local government vaccination campaign. It can also include patients that receive a third or fourth boost.
  Interventions: Drug: COVID-19 Vaccines
- Ad5-nCoV: Group of patients of any age, any sex, that will receive a complete scheme of approved Ad5-nCoV vaccination, assigned by a local government vaccination campaign. It can also include patients that receive a third or fourth boost.
  Interventions: Drug: COVID-19 Vaccines
- Gam-COVID-Vac: Group of patients of any age, any sex, that will receive a complete scheme of approved Gam-COVID-Vac vaccination, assigned by a local government vaccination campaign. It can also include patients that receive a third or fourth boost.
  Interventions: Drug: COVID-19 Vaccines
- Coronavac: Group of patients of any age, any sex, that will receive a complete scheme of approved Coronavac vaccination, assigned by a local government vaccination campaign. It can also include patients that receive a third or fourth boost.
  Interventions: Drug: COVID-19 Vaccines

INTERVENTIONS:
Drug: COVID-19 Vaccines — Each group will receive a complete scheme of the vaccine according to local government assignation

SUMMARY:
Background: Scarce information exists in relation to the comparison of seroconversion and adverse events following immunization (AEFI) with different SARS-COV2 vaccines. Our aim was to correlate the magnitude of the antibody response to vaccination with previous clinical conditions and AEFI.

Methods: A multicentric comparative study where SARS-CoV-2 spike 1-2 IgG antibodies IgG titers are being measured at baseline, 21-28 days after the first and second dose (when applicable), six months and a year of the following vaccines: BNT162b2 mRNA, mRNA-1273, Gam-COVID-Vac, Coronavac, ChAdOx1-S, Ad5-nCoV and Ad26.COV2. Mixed model and Poisson generalized linear models will be performed for the analyses.

DETAILED DESCRIPTION:
The aim of this study is to compare the seroconversion after the first and second dose (if applicable) between BNT162b2 mRNA, mRNA-1273, ChAdOx1-S, Ad26.COV2, Ad5-nCoV, Gam-COVID-Vac, and Coronavac through the measurement of SARS-CoV-2 spike 1-2 IgG antibodies using the same standardized assay.

Our secondary aims are to correlate the magnitude of the antibody response with previous clinical conditions (medical history) and previous diagnosis of SARS-CoV-2.

Our tertiary aim will be to compare the change in antibody levels after a third or fourth dose of any of the vaccines previously described

Also, we will investigate the differences across vaccines regarding adverse events after vaccination and determine the best predictors of systemic and severe adverse events.

This is a multicentric observational study of volunteers who will receive an approved complete scheme of BNT162b2 mRNA, mRNA-1273, ChAdOx1-S, Ad26.COV2, Ad5-nCoV, Gam-COVID-Vac, or Coronavac COVID-19 vaccine during 2021 in five hospital centers (Hospital Clinica Nova, Humanitas Clinical and Research Center, Fundación San Francisco Xavier, Ternium Health Center in Rio, Hospital Municipal San Jose, Hospital Interzonal de Agudos San Felipe) from four different countries: Mexico, Italy, Brazil and Argentina.

The study was approved by each local Institutional Review Board and conducted per the Code of Ethics of the World Medical Association (Declaration of Helsinki) for experiments that involve humans.

The inclusion criteria are: workers/participants of both genders at relevant vaccination places who consented to participate, planned to conclude the immunization regimen of any vaccine and agreed to be followed-up for the duration of the study. The following vaccines are available at sites at the time of the study: BNT162b2 mRNA, mRNA-1273, ChAdOx1-S, Ad26.COV2, Ad5-nCoV, Gam-COVID-Vac, or Coronavac. The exclusion criteria is to have been previously given any COVID-19 vaccine prior to study entry.

The vaccines available, the schedule of doses was defined by the Health System of each country, so that the day and the type of vaccine that each volunteer received has been assigned by the latter. At the vaccination day and prior to the vaccination, the research team invited any subject who planned to receive any scheme of vaccine.

The participant will recieve an explanation of the project and asked to sign the informed consent. Inclusion-exclusion criteria were applied and a plasma sample will be collected.

The baseline sample will be taken before receiving the first dose of any COVID-19 vaccine (T0). After 21 days (+/- 7 days) of the first dose, Then, 21 days (+/- 7 days) after the second dose (if applicable), six months, and a year after.

In case a patient receives a third or fourth dose of any vaccine, extra plasma samples for the antibody measures will be performed 21 days (+/- 7 days) after the third or fourth dose (if applicable), three months and six months after.

At each visit participants will have to answer a questionnaire.

The basal-sample questionnaire aimed at obtaining patients medical history and previous SARS-CoV-2 infections. The questionnaires will be applied after the first and second doses of vaccines to recognise adverse events and identify a potential SARS-CoV-2 infection after receiving any vaccine dose. SARS-CoV-2 infection will be also monitored by the epidemiology team through PCR test, which informed the research team of any new infection.

IgG determination To determine the amount of specific anti-S1 and anti-S2 IgG antibodies against SARS-CoV-2 in plasma samples, the laboratory personnel will use a chemiluminescence immunoassay (CLIA) developed by DiaSorin, which has a sensitivity of 97.4% (95% CI, 86.8-99.5) and a specificity of 98.5% (95% CI, 97.5-99.2). The results will be reported as follows: <12.0 AU / ml was considered negative, 12.0 to 15.0 AU / ml was indeterminate, and > 15 AU / ml was positive. This kit is comparable with other commercial kits such as Euroimmun and Roche, and has been used elsewhere.

The variables that will be analyzed are age, sex, personal medical history (for example the presence of type 2 diabetes, hypertension, asthma, pulmonary obstructive disease, any heart condition, obesity, cancer, liver steatosis, any autoimmune disease) including confirmed SARS-CoV-2 diagnosis (confirmed either with a nasal swab or serologic tests before and after vaccine shots), and adverse events after immunization (AEFI) caused by any dose of any vaccine. We will focuse on the following systemic or severe adverse events: fever (>37.5°C), adenopathy, diffuse rash, edema, facial paralysis, orthostatic hypotension, headache, arthralgia, myalgia, nausea, vomit and diarrhea. The analyzed biochemical variables are SARS-CoV-2 quantitative antibodies from baseline, 21-28 days post-first dose (S1), 21-28 days post-second dose if applicable, six and 12 months after vaccine application.

Statistical Methods The researchers will review the quality control and the anonymization of the database. Normality assumption will be evaluated with the Shapiro Wilk test, Kolmogorov and frequency histograms. Descriptive statistics such as mean, standard deviation, median, interquartile range, frequencies, and percentages will be computed. Mixed model and Poisson generalized linear models will be performed for analysis. A sample size of 1870 patients is calculated, according to the primary aim, by using a mixed model formula with an alpha of 0.05, power of 90%, the effect size of 0.15, and k=7. The analyses will be two-tailed. A p-value less than 0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Participants of both genders at relevant vaccination places who consented to participate, planned to conclude the immunization regimen of any vaccine and agree to be followed-up for the duration of the study

Exclusion Criteria:

* Previously given any SARS-CoV-2 vaccine prior to study entry

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study will include participants of both genders any age, that plan to receive a complete scheme of any of the next vaccines: BNT162b2 mRNA, mRNA-1273, ChAdOx1-S, Ad26.COV2, Ad5-nCoV, Gam-COVID-Vac, or Coronavac. From specified vaccination centres in Mexico, Brazil, Italy and Argentina
Sampling Method: Non-Probability Sample
Enrollment: 1870 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Seroconversion after first and second dose of SARS-COV2 vaccines | six months
  seroconversion after the first and second dose (if applicable) between BNT162b2 mRNA, mRNA-1273, ChAdOx1-S, Ad26.COV2, Ad5-nCoV, Gam-COVID-Vac, and Coronavac through the measurement of SARS-CoV-2 spike 1-2 IgG antibodies using the same standardized assay

SECONDARY OUTCOMES:
Adverse reaction after first and second dose of SARS-COV-2 vaccines | 6 months
  Determine differences across vaccines regarding adverse events after vaccination

OTHER OUTCOMES:
Seroconversion after third and fourth dose of SARS-Cov-2 vaccines | 6 months
  seroconversion after the third and fourth dose (if applicable) between BNT162b2 mRNA, mRNA-1273, ChAdOx1-S, Ad26.COV2, Ad5-nCoV, Gam-COVID-Vac, and Coronavac through the measurement of SARS-CoV-2 spike 1-2 IgG antibodies using the same standardized assay
Adverse reaction after third and fourth dose of SARS-COV-2 vaccines | 6 months
  Determine differences across vaccines regarding adverse events after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Maria Elena Romero-Ibarguengoitia, MD, MS, PHD, Principal Investigator — Hospital Clinica Nova de Monterrey
Locations (1):
- Hospital Clinica Nova de Monterrey, San Nicolás de los Garza, Mexico

IPD SHARING:
Plan to Share IPD: No
upon request

REFERENCES:
- [Derived] Romero-Ibarguengoitia ME, Gonzalez-Cantu A, Pozzi C, Levi R, Mollura M, Sarti R, Sanz-Sanchez MA, Rivera-Salinas D, Hernandez-Ruiz YG, Armendariz-Vazquez AG, Del Rio-Parra GF, Barco-Flores IA, Gonzalez-Facio R, Azzolini E, Barbieri R, de Azevedo Dias AR, Henriques Guimaraes Junior M, Bastos-Borges A, Acciardi C, Paez-Bo G, Teixeira MM, Rescigno M. Analysis of immunization time, amplitude, and adverse events of seven different vaccines against SARS-CoV-2 across four different countries. Front Immunol. 2022 Jul 28;13:894277. doi: 10.3389/fimmu.2022.894277. eCollection 2022. PMID 35967368